CLINICAL TRIAL: NCT02671877
Title: Preoperative Fibroscopy as a Predictor of the Difficulty of Laryngoscopy and Intubation
Acronym: TubeDiff
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Marco Gemma, Professor, MD, IRCCS San Raffaele
Other Study IDs: 132/ INT /2015
Record Dates: First submitted 2016-01-23; First posted 2016-02-02 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Tracheal Intubation Morbidity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Transnasal fiberoscopy — Minimally invasive exploration ot the upper airways, performed in an awake or minimally sedated patient.

SUMMARY:
The aim of this study is the evaluation of preoperative transnasal fiberoscopy, as a possible predictor of difficult laryngoscopy and intubation during elective general anesthesia in an adult population.

Transnasal fibercoscopy is a minimally invasive examination and is routinely performed during ENT evaluation; on the other hand, current strategies used to predict the ease of intubation are still not sufficiently sensitive and specific, and an unexpected difficult or failed intubation at the induction of general anesthesia is a seriuos, and potentially fatal, emergency in anesthesia.

In literature, a correlation between anatomical and functional parameters highlighted by fiberoscopy and difficulty of laryngoscopy and intubation has never been demonstrated nor indagated.

If proven, this might give the Anesthestiologist further information about the expected difficulty of laryngoscopy and intubation, guiding a different - and hopefully safer - anesthesiological strategy.

DETAILED DESCRIPTION:
This is a prospective, single-center, observational study. Aim of this study is the evaluation of preoperative transnasal fiberoscopy as a predictor of difficult laryngoscopy and intubation during elective general anesthesia in an adult population. Unexpected difficult of failed intubation is a serious, and potentially fatal, occurrence at the induction of general anesthesia. However, current strategies used to predict the ease of intubation are still not sufficiently sensitive and specific.

Patients undergoing a scheduled ENT (Ear-Nose-Throat) surgical intervention are subjected to a transnasal fibescopy, a minimally invasive examination, as a part of a normal ENT evaluation before surgery, according to the guidelines of the recruiting center.

During fiberoscopy, the investigators are collecting many anatomical and functional data about the upper airways of the patient. These data include the collapse of the upper airway during the Muller maneuver, the Cormack - Lehane scale as seen in fiberoscopy, the anatomy of the glottis and epiglottis.

The investigators are also collecting data about the preoperative evaluation made by the Anesthesiologist as well as the effective difficulty of laryngoscopy and intubation encountered at the induction of general anaesthesia, expressed by the Cormack - Lehane scale and the Intubation Difficulty Scale (IDS) as described in literature.

General anesthesia will be performed as usual and will not be influenced by fiberoptic evaluation as the Anesthesiologist will be blind to it, and he/she will be free to choose the best anesthesiological plan for his/her patient; whether an elective awake intubation will be chosen, this will exclude the patient from the study.

For safety reasons, the only exception to blindness is an expected difficulty of intubation > 90% (as reported in a VAS scale) by the ENT specialist, based upon the physician's experience. In this case, he will talk to the Anesthesiologist about and the patient will be excluded from the study.

The researchers are excluding from the study patients with suspect or confirmed malignancy of the nose, mouth, pharynx and larynx, as well as patients with trachoestomy, active bleeding lesions or those in which is planned an elective awake intubation for any reason.

To reduce confounders, the fiberoscopy will performed by an ENT specialist chosen in a limited pool (three) and it will be recorded and subsequently reviewed by another one in the same pool. Likewise, general anesthesia will be performed by a limited pool (three) of Anesthesiologists expert in ENT surgery.

Preoperative data obtained by fiberoscopy and intraoperative data recorded by the Anesthesiologist will be matched and analyzed, to explore a possibile relationship.

In literature, this relationship has never been demonstrated nor indagated. If proven, this might give the Anesthestiologist further information about the prediction of a difficult laryngoscopy and intubation, even beyond ENT surgery; in fact, whether fiberoscopy is routinely carried out for surgical reasons (e.g. vascular surgery for the evaluation of recurrent laryngeal nerve prior to aortic surgey) or requested by the Anesthesiologist him/herself at the moment of the preoperative evaluation, it might guide a different - and hopefully safer - anesthesiological strategy.

ELIGIBILITY:
Inclusion Criteria:

* Candidate to elective ENT surgery under general anesthesia

Exclusion Criteria:

* Subjects with suspect or ascertained malignancy of the nose, mouth, phayrx, or larynx that may interfere with tracheal intubation
* Subjects with tracheostomy
* Subjects with active bleeding or waiting for ENT surgery of bleeding lesions
* Subjects candidate to elective awake intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients candidate to elective Ear-Nose-Throat (ENT) surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2017-03-01 (Estimated)

PRIMARY OUTCOMES:
Difficulty of tracheal intubation | Intraoperative (single assessment)
  The difficulty of intubation is described with and the Intubation Difficulty Scale (IDS).

SECONDARY OUTCOMES:
Difficulty of tracheal laryngoscopy | Intraoperative (single assessment)
  The difficulty of tracheal laryngoscopy is described with the Cormack - Lehane Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Beretta Luigi, Full Professor, MD, Principal Investigator — IRCCS San Raffaele Hospital and San Raffaele University, Milan, Italy
Locations (1):
- S. Raffaele Hospital, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heinrich S, Birkholz T, Irouschek A, Ackermann A, Schmidt J. Incidences and predictors of difficult laryngoscopy in adult patients undergoing general anesthesia : a single-center analysis of 102,305 cases. J Anesth. 2013 Dec;27(6):815-21. doi: 10.1007/s00540-013-1650-4. Epub 2013 Jun 9. PMID 23748552
- [Background] Cormack RS, Lehane J. Difficult tracheal intubation in obstetrics. Anaesthesia. 1984 Nov;39(11):1105-11. PMID 6507827
- [Background] Adnet F, Borron SW, Racine SX, Clemessy JL, Fournier JL, Plaisance P, Lapandry C. The intubation difficulty scale (IDS): proposal and evaluation of a new score characterizing the complexity of endotracheal intubation. Anesthesiology. 1997 Dec;87(6):1290-7. doi: 10.1097/00000542-199712000-00005. PMID 9416711
- [Background] Vannucci A, Cavallone LF. Bedside predictors of difficult intubation: a systematic review. Minerva Anestesiol. 2016 Jan;82(1):69-83. Epub 2015 May 20. PMID 25990431
- [Derived] Gemma M, Buratti L, Di Santo D, Calvi MR, Ravizza A, Bondi S, Bussi M, Beretta L. Pre-operative transnasal endoscopy as a predictor of difficult airway: A prospective cohort study. Eur J Anaesthesiol. 2020 Feb;37(2):98-104. doi: 10.1097/EJA.0000000000001127. PMID 31789897